CLINICAL TRIAL: NCT05844254
Title: Patient Centered Outcomes and Stability of Root Coverage by Novel Overlapping Rotated Double (NORD) Flap as Compared to Sub Epithelial Connective Tissue Graft in Isolated Recession type1 Gingival Recession-A Randomized Controlled Trial
Brief Title: Comparison of Root Coverage Outcomes by NORD Flap Versus Subepithelial Connective Tissue Graft in RT1 Gingival Recession
Acronym: Recession type
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr. Ritika Arora perio 2023
Record Dates: First submitted 2023-02-01; First posted 2023-05-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Gingival Recession
Keywords: Sub epithelial connective tissue graft; patient centered outcomes; phenotype
MeSH Terms: conditions — Gingival Recession | interventions — Surgical Flaps

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NORD group (Experimental): After undergoing phase one of periodontal therapy, patients will be recalled after four weeks for root coverage surgery. NORD group will undergo NORD flap for root coverage. Patients will be followed up after 1 month,6, 12 and 15 months. Patients belonging to thin phenotype will be followed up as separate cohort for period of one year to evaluate phenotype modification.
  Interventions: Procedure: novel overlapping rotated double (NORD) flap
- Sub epithelial connective tissue group (Active Comparator): After undergoing phase one of periodontal therapy, patients will be recalled after four weeks for root coverage surgery. Sub epithelial connective tissue group will receive sub epithelial connective tissue graft. Patients will be followed up after 1 month,6, 12 and 15 months. Patients belonging to thin phenotype will be followed up as separate cohort for period of one year to evaluate phenotype modification.
  Interventions: Procedure: novel overlapping rotated double (NORD) flap

INTERVENTIONS:
Procedure: novel overlapping rotated double (NORD) flap — After undergoing phase one of periodontal therapy, patients will be recalled after four weeks for root coverage surgery. Patients will be randomly allotted to either group by stratified block randomization after taking baseline measurement with respect to periodontal phenotype(PP) [using transparency of periodontal probe through the gingival margin, when probe is visible, thin PP and when not visible, thick PP] so that patients with thick and thin PP get an equal chance of being allocated to NORD and Sub epithelial connective tissue group.
  1. Group 1(NORD group)- Patients treated with NORD flap
  2. Group 2 (Sub epithelial connective tissue group)- Patients treated with sub epithelial connective tissue graft Patients will be followed up after 1 month,6, 12 and 15 months. 30 patients belonging to thin phenotype will be followed up as separate cohort for period of one year to evaluate phenotype modification.

SUMMARY:
Management of GR in the initial stages (when there is no inter proximal attachment and bone loss involved) has better clinical outcomes and reduces the chances of further progression of recession. Surgical treatment of recession involves techniques like pedicle grafts and free soft tissue grafts and their modifications. Sub epithelial connective tissue graft is considered as the gold standard in root coverage techniques. However this procedure involves a second surgical site increasing surgical time, complexity and patient morbidity. So there is a need of a technique which overcomes these limitations, is easier to perform and helps to achieve comparable root coverage with stable results over a long term. Novel overlapping rotated double (NORD) flap is a novel technique which offers a solution to this problem. This may help to achieve greater thickness of gingiva in the region of GR after healing and may reduce the risk of future recession. This technique is being compared with the bilaminar technique utilizing the sub epithelial connective tissue graft at the control sites, both the test and control groups will be treated using a microsurgical approach. If there is no significant difference in the root coverage achieved between the two techniques, this may reduce the need of harvesting connective tissue graft from a second surgical site. This

technique is also expected to have better patient reported outcomes and will benefit the patients and operator both. This technique may also help to modify the phenotype of the affected tooth, thus making the results more stable.

DETAILED DESCRIPTION:
Gingival recession (GR) is a very frequent finding in the general population with a prevalence ranging from 50-90% in different populations. Patients with GR may experience hypersensitivity, pain, poor esthetics and difficulty in maintaining oral hygiene. Among the predisposing factors for GR, most common are improper tooth brushing, gingival inflammation, thin periodontal phenotype, aberrant frenum, areas with inadequate keratinized gingiva, orthodontic movement leading to buccal tooth displacement and direct trauma. Literature suggests that untreated gingival recession has a high probability of undergoing further progression even in the presence of good oral hygiene. From an epidemiological point of view, localized facial gingival recessions affect more than 60% of individuals and account for a significant amount of periodontal attachment loss in subjects with good oral hygiene; therefore there is a need for predictable root coverage techniques. Many surgical techniques have been shown to be effective in correcting gingival recession by covering the exposed root with soft tissue; however, the thickness of the gingival tissue over the root surface probably plays an important role in preventing the recurrence of tissue recession. To cover the exposed root surfaces numerous techniques with various modifications have been attempted with the main focus in the recent decades being on complete root coverage. Pedicle grafts are usually considered superior to free soft tissue grafts due to intact blood supply from the donor site. Laterally positioned flap and double papilla grafts are examples of pedicle grafting techniques that obtain advantage of available keratinized tissue from the neighboring teeth. However, there is a risk of developing recession on the donor tooth or in case of double papilla flap, an inadequate coverage due to wound edges being sutured over an avascular surface. This is especially important in cases of thin periodontal phenotype. Sub epithelial connective tissue graft, though considered as a gold standard among the soft tissue grafting techniques involves a second surgical site increasing surgical time, complexity and patient morbidity. . To overcome these limitations, a novel technique is being proposed here.

9. Methodology

i. Study design- This randomized controlled trial will be conducted in the department of Periodontics, Post graduate institute of dental sciences (PGIDS), Rohtak in accordance with the ethical standards outlined in the declaration of Helsinki 1975, as revised in 2013.The study design was approved by Institutional review board, PGIDS, Rohtak and ethical acceptance applied for from the Ethical committee of PGIDS, Rohtak.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18-45 years

  * Non smokers (current and past smokers
  * Plaque index ≤1,Gingival index≤1
  * RT1(Miller's class I and class II)gingival recession, that is, GR with no loss of inter proximal attachment
  * Probing depth ≤3 mm
  * Width of attached gingiva≥3 mm on the mesial and distal sides of the recipient tooth.
  * Adequate vestibular depth

Exclusion Criteria:

* • Patients with a history of any systemic condition that might alter the course of disease and

  * or wound healing such as diabetes mellitus, immunologic disorders, cardio-vascular disease etc.

    * Pregnant and lactating women.
    * Patients with immature tooth.
    * Patients with tooth fracture or tooth mobility
    * Patients receiving treatment with antibiotics, statins, glucocorticoids, bisphosphonates or any other modulatory drug.
    * Patients undergoing orthodontic treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-02 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Recession depth | 1month
  change in recession depth from baseline at 1month will be assessed. The unit of measurement is millimeter.
Change in Recession depth | 6months
  change in recession depth from baseline at 6months will be assessed. The unit of measurement is millimeter.
Change in Recession depth | 12months
  change in recession depth from baseline at 12months will be assessed. The unit of measurement is millimeter.
Change in Recession depth | 15months
  change in recession depth from baseline at 15months will be assessed. The unit of measurement is millimeter.
Root coverage (%)- Change in recession depth/RD at baseline × 100 | 1month
  change in recession depth from baseline to 1month will be assessed. The obtained value would be divided by recession depth at baseline. The value obtained would be multiplied by 100. The unit of measurement is millimeters.
Root coverage (%)- change in recession depth/RD at baseline × 100 | 6 months
  change in recession depth from baseline to 6months will be assessed. The obtained value would be divided by recession depth at baseline. The value obtained would be multiplied by 100. The unit of measurement is millimeters.
Root coverage (%)-Change in recession depth/RD at baseline × 100 | 12months
  change in recession depth from baseline to 12months will be assessed. The obtained value would be divided by recession depth at baseline. The value obtained would be multiplied by 100. The unit of measurement is millimeters.
Root coverage (%)- change in recession depth/RD at baseline × 100 | 15months
  change in recession depth from baseline to 15months will be assessed. The obtained value would be divided by recession depth at baseline. The value obtained would be multiplied by 100. The unit of measurement is millimeters.
Visual analog scale | 24 hours after surgery
  Patients will be asked to record their pain using Visual analog scale (VAS) from 0 to 100, with 0 representing no pain and 100 representing pain as bad as it could be.
Visual analog scale | 10 days after surgery
  Patients will be asked to record their pain using Visual analog scale (VAS) from 0 to 100, with 0 representing no pain and 100 representing pain as bad as it could be.
Visual analog scale | 1month
  Patients will be asked to record their pain using Visual analog scale (VAS) from 0 to 100, with 0 representing no pain and 100 representing pain as bad as it could be.
Visual analog scale | 6months
  Patients will be asked to record their pain using Visual analog scale (VAS) from 0 to 100, with 0 representing no pain and 100 representing pain as bad as it could be.
Visual analog scale | 12 months
  Patients will be asked to record their pain using Visual analog scale (VAS) from 0 to 100, with 0 representing no pain and 100 representing pain as bad as it could be.
Visual analog scale | 15 months
  Patients will be asked to record their pain using Visual analog scale (VAS) from 0 to 100, with 0 representing no pain and 100 representing pain as bad as it could be.
Patient centered outcomes | 10 days after surgery
  All Patient centered outcomes would be recorded in the questionnaire
Patient centered outcomes | 1month
  All Patient centered outcomes would be recorded in the questionnaire

SECONDARY OUTCOMES:
Probing depth | baseline
  Probing depth (in millimeter) would be measured from gingival margin to the base of pocket at six sites per tooth.
Probing depth | 1month
  Probing depth (in millimeter) would be measured from gingival margin to the base of pocket at six sites per tooth.
Probing depth | 6 months
  Probing depth (in millimeter) would be measured from gingival margin to the base of pocket at six sites per tooth.
Probing depth | 12 months
  Probing depth (in millimeter) would be measured from gingival margin to the base of pocket at six sites per tooth.
Probing depth | 15 months
  Probing depth (in millimeter) would be measured from gingival margin to the base of pocket at six sites per tooth.
Clinical attachment level | baseline
  Probing depth (in millimeter) would be measured from cemento-enamel junction to base of the pocket at six sites per tooth.
Clinical attachment level | 1month
  Probing depth (in millimeter) would be measured from cemento-enamel junction to base of the pocket at six sites per tooth.
Clinical attachment level | 6 months
  Probing depth (in millimeter) would be measured from cemento-enamel junction to base of the pocket at six sites per tooth.
Clinical attachment level | 12 months
  Probing depth (in millimeter) would be measured from cemento-enamel junction to base of the pocket at six sites per tooth.
Clinical attachment level | 15 months
  Probing depth (in millimeter) would be measured from cemento-enamel junction to base of the pocket at six sites per tooth.
Recession depth- at recipient tooth only | baseline
  recession depth (in millimeter) would be measured as a distance from the cemento-enamel junction to the most apical point of the buccal gingival margin
Recession depth- at recipient tooth only | 1month
  recession depth (in millimeter) would be measured as a distance from the cemento-enamel junction to the most apical point of the buccal gingival margin
Recession depth- at recipient tooth only | 6months
  recession depth (in millimeter) would be measured as a distance from the cemento-enamel junction to the most apical point of the buccal gingival margin
Recession depth- at recipient tooth only | 12months
  recession depth (in millimeter) would be measured as a distance from the cemento-enamel junction to the most apical point of the buccal gingival margin
Recession depth- at recipient tooth only | 15months
  recession depth (in millimeter) would be measured as a distance from the cemento-enamel junction to the most apical point of the buccal gingival margin
Recession width- at recipient tooth only | baseline
  recession width (in millimeter) would be measured by placing the periodontal probe horizontally at the most apical point of buccal cemento-enamel junction. The distance from the gingival margin mesial to a point distal of the recession will be measured.
Recession width- at recipient tooth only | 1month
  recession width (in millimeter) would be measured by placing the periodontal probe horizontally at the most apical point of buccal cemento-enamel junction. The distance from the gingival margin mesial to a point distal of the recession will be measured.
Recession width- at recipient tooth only | 6months
  recession width (in millimeter) would be measured by placing the periodontal probe horizontally at the most apical point of buccal cemento-enamel junction. The distance from the gingival margin mesial to a point distal of the recession will be measured.
Recession width- at recipient tooth only | 12months
  recession width (in millimeter) would be measured by placing the periodontal probe horizontally at the most apical point of buccal cemento-enamel junction. The distance from the gingival margin mesial to a point distal of the recession will be measured.
Recession width- at recipient tooth only | 15months
  recession width (in millimeter) would be measured by placing the periodontal probe horizontally at the most apical point of buccal cemento-enamel junction. The distance from the gingival margin mesial to a point distal of the recession will be measured.
width of keratinised gingiva | baseline
  Distance would be measured from gingival margin to muco-gingival junction at mid-buccal site to calculate width of keratinized gingiva. From the calculated width of keratinized gingiva, subtract the Probing depth at mid-buccal site.
Width of keratinised gingiva | 1month
  Distance would be measured from gingival margin to muco-gingival junction at mid-buccal site to calculate width of keratinized gingiva. From the calculated width of keratinized gingiva, subtract the Probing depth at mid-buccal site.
Width of keratinised gingiva | 6months
  Distance would be measured from gingival margin to muco-gingival junction at mid-buccal site to calculate width of keratinized gingiva. From the calculated width of keratinized gingiva, subtract the Probing depth at mid-buccal site.
Width of keratinised gingiva | 12months
  Distance would be measured from gingival margin to muco-gingival junction at mid-buccal site to calculate width of keratinized gingiva. From the calculated width of keratinized gingiva, subtract the Probing depth at mid-buccal site.
Width of keratinised gingiva | 15months
  Distance would be measured from gingival margin to muco-gingival junction at mid-buccal site to calculate width of keratinized gingiva. From the calculated width of keratinized gingiva, subtract the Probing depth at mid-buccal site.
Gingival thickness | baseline
  Gingival thickness will be measured 1.0mm apical to gingival margin using an injection needle, perpendicular to tissue surface, and a silicon stop over gingival surface. The silicon disc stop will be placed in tight contact with soft tissue. After needle removal, the distance between needle tip and silicon stop will be estimated using a digital caliper with 0.01mm of accuracy.
Gingival thickness | 1month
  Gingival thickness will be measured 1.0mm apical to gingival margin using an injection needle, perpendicular to tissue surface, and a silicon stop over gingival surface. The silicon disc stop will be placed in tight contact with soft tissue. After needle removal, the distance between needle tip and silicon stop will be estimated using a digital caliper with 0.01mm of accuracy.
Gingival thickness | 6 months
  Gingival thickness will be measured 1.0mm apical to gingival margin using an injection needle, perpendicular to tissue surface, and a silicon stop over gingival surface. The silicon disc stop will be placed in tight contact with soft tissue. After needle removal, the distance between needle tip and silicon stop will be estimated using a digital caliper with 0.01mm of accuracy.
Gingival thickness | 12 months
  Gingival thickness will be measured 1.0mm apical to gingival margin using an injection needle, perpendicular to tissue surface, and a silicon stop over gingival surface. The silicon disc stop will be placed in tight contact with soft tissue. After needle removal, the distance between needle tip and silicon stop will be estimated using a digital caliper with 0.01mm of accuracy.
Gingival thickness | 15 months
  Gingival thickness will be measured 1.0mm apical to gingival margin using an injection needle, perpendicular to tissue surface, and a silicon stop over gingival surface. The silicon disc stop will be placed in tight contact with soft tissue. After needle removal, the distance between needle tip and silicon stop will be estimated using a digital caliper with 0.01mm of accuracy.
Change in Recession width | 1month
  Change in recession width would be measured from baseline to 1month.
Change in Recession width | 6 months
  Change in recession width would be measured from baseline to 6months.
Change in Recession width | 12 months
  Change in recession width would be measured from baseline to 12months.
Change in Recession width | 15 months
  Change in recession width would be measured from baseline to 15months.
Root coverage-esthetic score | 1month
  According to Root coverage-esthetic score system 5 variables will be assessed. The variables are: level of gingival margin, marginal tissue contour, soft tissue texture, muco-gingival junction alignment, gingival colour.
  A score of 0,3, or 6 will be used for the evaluation of gingival margin position, whereas a score of 0-1 will be used for each of the other variables. The highest and best aesthetic score to be achieved for complete root coverage is 10.
Root coverage-esthetic score | 6 months
  According to Root coverage-esthetic score system 5 variables will be assessed. The variables are: level of gingival margin, marginal tissue contour, soft tissue texture, muco-gingival junction alignment, gingival colour.
  A score of 0,3, or 6 will be used for the evaluation of gingival margin position, whereas a score of 0-1 will be used for each of the other variables. The highest and best aesthetic score to be achieved for complete root coverage is 10.
Root coverage-esthetic score | 12 months
  According to Root coverage-esthetic score system 5 variables will be assessed. The variables are: level of gingival margin, marginal tissue contour, soft tissue texture, muco-gingival junction alignment, gingival colour.
  A score of 0,3, or 6 will be used for the evaluation of gingival margin position, whereas a score of 0-1 will be used for each of the other variables. The highest and best aesthetic score to be achieved for complete root coverage is 10.
Root coverage-esthetic score | 15 months
  According to Root coverage-esthetic score system 5 variables will be assessed. The variables are: level of gingival margin, marginal tissue contour, soft tissue texture, muco-gingival junction alignment, gingival colour.
  A score of 0,3, or 6 will be used for the evaluation of gingival margin position, whereas a score of 0-1 will be used for each of the other variables. The highest and best aesthetic score to be achieved for complete root coverage is 10.

CONTACTS AND LOCATIONS:
Overall Officials: RITIKA ARORA, M.D.S., Principal Investigator — Post Graduate Institute of Dental Sciences, Rohtak
Locations (1):
- Post graduate institute of dental sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No